CLINICAL TRIAL: NCT01043211
Title: Analgesic Efficacy of Intravenous Lidocaine for Postoperative Pain Following Adult Spine Surgery: A Randomized Controlled Trial
Brief Title: Analgesic Efficacy of Intravenous Lidocaine for Postoperative Pain Following Adult Spine Surgery
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Did not have the research staff necessary to follow through with this study.
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: F091105002
Record Dates: First submitted 2009-12-28; First posted 2010-01-06 (Estimated); Last update posted 2015-03-10 (Estimated); Status verified 2015-01

CONDITIONS: Back Pain
Keywords: Back Pain; Lidocaine
MeSH Terms: conditions — Back Pain | interventions — Lidocaine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Lidocaine Hydrochoride Injection, without epinephrine — A standardized 0.2 ml/kg (2 mg/kg) intravenous bolus dose of lidocaine (1%, 10 mg/ml) is given after anesthetic induction but prior to skin incision. Immediately thereafter, lidocaine (1%, 10 mg/ml) will be administered on a standardized 0.3 ml/hr/kg (3 mg/kg/hr, maximum 200 mg/hr = 20 ml/hr) basis using a continuous infusion pump during the surgical procedure. Immediately after skin closure, the lidocaine infusion will be decreased by 50% to 0.15 ml/hr/kg (1.5 mg/kg/hr, maximum 100 mg/hr = 10 ml/hr) and continued for 90 minutes postoperatively. The infusion will be stopped before the patient is discharged from the post-anesthesia care unit (PACU).
  Other Names: Xylocaine
Drug: Normal Saline — A standardized 0.2 ml/kg intravenous bolus dose of preservative-free normal saline will be given after anesthetic induction but prior to skin incision. Immediately thereafter, normal saline will be administered on an equal 0.3 ml/hr/kg (maximum 20 ml/hr) basis using a continuous infusion pump during the surgical procedure. Immediately after skin closure, the normal saline infusion will be decreased by 50% to 0.15 ml/hr/kg (maximum 10 ml/hr) and continued for 90 minutes postoperatively. The infusion will be stopped before the patient is discharged from the post-anesthesia care unit (PACU).
Drug: Normal Saline — A standardized 0.2 ml/kg (2 mg/kg) intravenous bolus dose of lidocaine (1%, 10 mg/ml) is given after anesthetic induction but prior to skin incision.

SUMMARY:
The purpose of this study is to generate further insight into the role and effectiveness of the amide local anesthetic lidocaine as an adjuvant postoperative analgesic after adult spine surgery. The effect of perioperative intravenous lidocaine infusion on postoperative rehabilitation and the inflammatory response will also be examined.

DETAILED DESCRIPTION:
Inadequate pain control after spine surgery in adults can result in increased patient morbidity and length of hospital stay, whereas improved postoperative pain control has been demonstrated to have numerous physiologic benefits and to reduce postoperative complications. When administered systemically, the amide local anesthetic lidocaine has potent anti-inflammatory properties, including inhibition of the arachidonic acid cascade and production of eicosanoids and prostaglandins. Previous studies have confirmed that the continuous intravenous administration of lidocaine during and after abdominal surgery in adults improves patient rehabilitation (specifically, pain intensity, duration of ileus, incidence of nausea and vomiting), and shortens hospital stay. The beneficial anti-inflammatory properties versus untoward side effects of the local anesthetics appear superior to steroids and the non-steroidal anti-inflammatory drugs (NSAIDs). Moreover, concern and controversy exists regarding the adverse effects of NSAIDs on bone healing, particularly in adults undergoing spine surgery.

No study to date has investigated the efficacy of a continuous perioperative lidocaine infusion in the adult spine surgery population. Therefore, in this prospective, randomized, controlled trial, we will evaluate the analgesic efficacy, anti-inflammatory properties, and rehabilitation pattern with a continuous, perioperative intravenous infusion of lidocaine versus a normal saline placebo in adult patients undergoing a decompressive lumbar laminectomy for spinal canal stenosis. Subjects enrolled in this study will receive a standardized general anesthetic that is consistent with our present clinical practice. The study participants will be randomized to receive both a perioperative bolus (2 mg/kg) and subsequent intravenous infusion (3 mg/kg/hr) of the amide local anesthetic lidocaine or a normal saline placebo at an equal volume per hour. The study infusion will be continued for 90 minutes after surgery. All patients will receive ample and adequate intravenous doses of an opioid (morphine sulfate) to reduce their pain intensity to acceptable levels. Pain intensity, opioid requirements, opioid-related side effects, and both the immediate and sustained rehabilitation pattern will be assessed. In addition to plasma lidocaine levels in the active drug group, plasma C-reactive protein, cortisol, and cytokine levels (e.g., IL-6, IL-10 and TNF-α) will be obtained at a series of perioperative time points in all study patients. Postoperative cytokine levels will also be measured in the surgical drainage fluid.

ELIGIBILITY:
Inclusion Criteria:

1. 19 years to 80 years of age
2. American Society of Anesthesiologists 1-3 status
3. Undergoing lumbar laminectomy between levels L1 and S1 for decompression of degenerative lumbar canal stenosis but without fusion or internal fixation performed

Exclusion Criteria:

1. American Society of Anesthesiologists 4 status
2. Previous spinal fusion surgery but patient may have undergone previous lumbar laminectomy or lumbar open discectomy
3. Morbid obesity (BMI > 40)
4. Diagnosis of spinal metastatic cancer
5. Presence of a severe or systemic bacterial infection
6. Allergy to an amide local anesthetic or morphine sulfate
7. History of a seizure disorder
8. History of atrial or ventricular arrhythmia
9. History of autonomic dysfunction (e.g., dysautonomia of diabetes)
10. History of renal dysfunction, liver dysfunction or congestive heart failure
11. History of substance abuse disorder
12. History of major psychiatric disorder (e.g., depression, bipolar disorder, Axis II personality disorder, schizophrenia)
13. Chronic opioid use of greater than 100 mg/day of morphine equivalents within 30 days prior to surgery
14. Current use of a corticosteroid
15. Use of a non-steroidal anti-inflammatory drug (NSAID), including low dose aspirin within the past 5 days
16. Use of an arrhythmic drug within the past 7 days
17. Current administration of a known potent CYP1A2 inhibitor, including zileuton (Zyflo), ciprofloxacin, enoxacin or any other fluoroquinolone antibiotic, amiodarone, mexiletine, propafenone, verapamil, cimetidine (Tagamet), famotidine (Pepcid), oral contraceptives, acyclovir (Zovirax) and ticlopidine (Ticlid) (Horn & Hansten, 2008).
18. Current administration of a known potent CYP3A4 inhibitor, including erythromycin, clarithromycin, azole antifungal (ketoconazole, fluconazole), verapamil, diltiazem, and grapefruit juice (Scuderi et al., 2006).
19. Pregnant females

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-01; Primary Completion 2013-12 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Postanesthesia care unit(PACU)admission duration (in minutes) | Assessed after discharge from PACU
Post extubation requirement for intravenous fentanyl in operating room (Y/N and mcg/kg) | Post extubation
Time to first nurse administered morphine dose after PACU admission (in minutes) | Assessed after PACU admission
Total dose of fentanyl administered intraoperatively (mcg/kg) and in the PACU (mcg/kg) | Measured post op
Total amount of mophine administered/PCA pump demands and doses and ratio of PCA demands/doses | 48-72 hours postoperative period
Self reported VAS pain scores (on a 0-100 scale) | Obtained on admissions to and upon discharge from PCAU, every 4 hours thereafter for the first 48 to 72 hours postoperatively, and at time of initial postoperative mobilization

SECONDARY OUTCOMES:
Side effect analysis | Measurements of side effect analysis will be done postoperatively
Pain Intensity Questionnaires | BPI-SF completed at time of initial and subsequent postop visits, Roland Morris Back Pain Questionnaire completed postop and 12-14 days, 3 mos, 6 mos, 12 mos, and 24 mos postop as compared to baseline value
Length of hospital stay | From admission to discharge
Post rehab analysis | Time to first liquid oral intake, time to initial mobilization, time to discontinuation of study solution infusion, time to discharge order, and to time to actual discharge home

CONTACTS AND LOCATIONS:
Overall Officials: Thomas R Vetter, M.D., M.P.H, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States